CLINICAL TRIAL: NCT04315168
Title: Evaluation of Safety and Efficacy of the FRED and FRED JR Devices for Intracranial Aneurysm Treatment
Brief Title: FRED and FRED JR Devices for Intracranial Aneurysm Treatment
Status: Completed | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FRED-EPI
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Intracranial Aneurysm
Keywords: aneurysm; endovascular; flow-diverter
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: FRED and FRED JR — Intracranial aneurysm treatment
  Other Names: Flow Re-Direction Endoluminal Device

SUMMARY:
A French, multicenter, prospective, observational, "real-world" assessment of the safety and efficacy of FRED and FRED Jr devices in the treatment of intracranial aneurysms

DETAILED DESCRIPTION:
Post Market Clinical Follow-up. Multicenter observational study. Treatment and follow-up far at least 12 months as per standard of care.

Sample Size: 138 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an intracranial aneurysm for which an endovascular treatment is indicated with the device FRED or FRED JR
* Patient or patient's legally authorized representative has been informed about the study and does not oppose the collection of his/her personal data

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with an intracranial aneurysm treated with the FRED or FRED JR Device
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality Rate | 1 year
  Percentage of patients with neurological death
Morbidity Rate | 1 year
  Percentage of patients with major ipsilateral stroke

SECONDARY OUTCOMES:
modified Rankin Score | 1 year
  worsening mRS (scale from 0 to 6 : 0= No symptom, 6= Death)
Complete aneurysm occlusion rate | 1 year
  Measured by the Raymond Scale
Retreatment Rate | 1 year
  Rate and description of aneurysm retreated or planned for retreatment
Patient description | 1 year
  Description of the population of patients treated with FRED and FRED JR in France

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Pierot, Prof., Principal Investigator — Hôpital Maison Blanche, Reims, France
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No